CLINICAL TRIAL: NCT04674878
Title: Comparison of Muscle Energy Techniques (METS) With Breathing Exercises to Improve Functional Outcomes in Patients of Fibromyalgia.
Brief Title: Comparison of Muscle Energy Techniques and Breathing Exercises for Functional Improvement in Fibromyalgia
Acronym: MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00705 Saira Zahid
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Fibromyalgia
Keywords: Diaphragmatic breathing; Fibromyalgia; Muscle energy techniques; Breathing exercises
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET group (Experimental): METs for accessory muscles of respiration including sternocleidomastoid, scalenes and trapezius given thrice a week for 8 weeks.
  Interventions: Other: METs
- Breathing exercise group (Active Comparator): Diaphragmatic breathing, pursed lip breathing and diaphragmatic breathing with resistance given thrice a week for 8 weeks.
  Interventions: Other: Breathing exercise group

INTERVENTIONS:
Other: METs — The isometric contraction of 7 sec will be applied followed by a stretching of 30 sec in painless range. This treatment will be given to the both sides of the neck targeting the three major accessory muscles of respiration.
  Arms: MET group
Other: Breathing exercise group — Three exercises will be performed in a circuit, 2 circuits in every session. It will include diaphragmatic breathing exercise in which patient will be in supine position inhaling through nose and expiration through moth with half closed lips. Second exercise pursed lip breathing also in supine position with the hands on abdomen and then inspiration through nose and expiration through mouth with half closing of lips. Third exercise resisted diaphragmatic breathing also in same pattern as second exercise with an addition of 1 kg weight on abdomen.
  Arms: Breathing exercise group

SUMMARY:
This study is planned to compare the effects of Muscle Energy Techniques (MET) with breathing exercises for improving functional outcomes in patients with fibromyalgia. A randomized controlled trial will be conducted. Sample size would be 26 patients with fibromyalgia randomly allocated to the Muscle energy techniques group and breathing exercise group. Both the groups will receive 8 weeks of treatment, 3 times per week. Data will be collected at baseline 5th week and 8th week. Outcome measurements include a Numeric pain rating scale, 6 min walk test, chest expansion, Pittsburgh sleep quality index, and Fibromyalgia Impact Questionnaire scores.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a common syndrome characterized by widespread pain and at least 11/18 painful tender points (American College of Rheumatology). Fibromyalgia syndrome (FMS) is a rheumatic condition of increasing prevalence worldwide) approximately 2-7% of the populations are affected. Some of the symptoms associated with fibromyalgia is sleep disturbance, dizziness, headache, fatigue, depression/tension, pain, cognitive disorder, irritable bowel syndrome, and different somatic symptoms. These factors negatively influence physical and emotional characteristics and decrease the quality of life. Fatigue and dyspnea are the significant signs and symptoms of fibromyalgia, which can be related to respiratory system changes. Major affected areas in fibromyalgia include breathing mechanics, the upper trapezius muscle, the cervical muscle mass, the scalene, Sternocleidomastoid, and the area around the second rib and all the paravertebral muscle mass. These regions are coordinated with the tender points placed in the upper half body of patients with FM. Fibromyalgia patients, without a doubt, exhaust and come to be fatigue due to the dyspnea. It is widespread among females; however, it can additionally affect both men and teenagers. Many pharmacological therapies were being used to treat FM with uncertain consequences, and steadily growing small doses are usually recommended to maximize efficacy. Among non pharmacological management including exercise is typically endorsed in the management of patients with fibromyalgia. Regular workout is an essential keystone of fibromyalgia management. Aerobic workout interventions have shown reduced ache, depression, and fatigue, improving health-related quality of life (HRQOL). Related literature includes meta-analysis regarding the exercise effects (endurance, aerobic, or mixed aerobic and strength workout) on worldwide welfare in people with fibromyalgia. Breathing issues tend to intensify FM symptoms. The FM patients exhaust quickly, and dyspnea causes fatigue related to respiratory muscle weakness, mainly diaphragmatic deficiency, that can decrease the physical condition and capability inside the daily activities. Breathing exercises have been proven to be useful in decreasing symptoms of FM. MET is the osteopathic manipulation strategies of the tender tissues that evolved to recover the musculoskeletal system's function and decrease pain. Both these techniques have proven effects for reduction of symptoms in FM patients. This study is intended to compare the effects of both in order to find out the technique that can effectively improve the functional outcomes in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology's criteria of fibromyalgia will be used

Exclusion Criteria:

* Smokers
* Severe spinal injuries
* Inflammatory rheumatic disease
* Patients diagnosed with pulmonary Disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale for pain (NPRS) | 8 weeks
  The Numeric Pain Rating Scale is a subjective measure, in which individuals rate their pain on an eleven point numeric scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Fibromyalgia impact questionnaire (FIQ) | 4 and 8 weeks
  The Fibromyalgia Impact Questionnaire is an assessment and evaluation instrument developed to measure fibromyalgia patient status, progress and functional capacity. It has been designed to measure the components of health status that are believed to be the most affected by FM.
6 Minute walk test (6MWT) | 4 and 8 weeks
  The 6-min walk test is a submaximal exercise test that entails measurement of distance walk over a span of 6 min. The 6-minute walk distance provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Pittsburgh sleep Quality Index (PSQI) | 4 and 8 weeks
  The Pittsburgh Sleep Quality Index is a self-report questionnaire assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produces one global score and takes 5-10 minutes to complete.
Measuring tape for the thoracoabdominal mobility indices | 4 and 8 weeks
  Measuring tape is used to measure thoracoabdominal expansion at three levels which are Axilla, Xiphoid and Navel.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Background] Forti M, Zamuner AR, Andrade CP, Silva E. Lung Function, Respiratory Muscle Strength, and Thoracoabdominal Mobility in Women With Fibromyalgia Syndrome. Respir Care. 2016 Oct;61(10):1384-90. doi: 10.4187/respcare.04401. Epub 2016 Apr 19. PMID 27094397
- [Background] Imamura M, Cassius DA, Fregni F. Fibromyalgia: From treatment to rehabilitation. Eur J Pain. 2009 Nov 1;3(2):117-122. doi: 10.1016/j.eujps.2009.08.011. PMID 20657807
- [Background] Sim J, Adams N. Systematic review of randomized controlled trials of nonpharmacological interventions for fibromyalgia. Clin J Pain. 2002 Sep-Oct;18(5):324-36. doi: 10.1097/00002508-200209000-00008. PMID 12218504
- [Background] Sarzi-Puttini P, Atzeni F, Salaffi F, Cazzola M, Benucci M, Mease PJ. Multidisciplinary approach to fibromyalgia: what is the teaching? Best Pract Res Clin Rheumatol. 2011 Apr;25(2):311-9. doi: 10.1016/j.berh.2011.03.001. PMID 22094204
- [Background] Garrido M, Castano MY, Biehl-Printes C, Gomez MA, Branco JC, Tomas-Carus P, Rodriguez AB. Effects of a respiratory functional training program on pain and sleep quality in patients with fibromyalgia: A pilot study. Complement Ther Clin Pract. 2017 Aug;28:116-121. doi: 10.1016/j.ctcp.2017.05.013. Epub 2017 May 28. PMID 28779918
- [Background] Tomas-Carus P, Branco JC, Raimundo A, Parraca JA, Batalha N, Biehl-Printes C. Breathing Exercises Must Be a Real and Effective Intervention to Consider in Women with Fibromyalgia: A Pilot Randomized Controlled Trial. J Altern Complement Med. 2018 Aug;24(8):825-832. doi: 10.1089/acm.2017.0335. Epub 2018 Apr 13. PMID 29653069